CLINICAL TRIAL: NCT02465528
Title: A Phase II, Open Label, Multi-center, Multi-arm Study of Ceritinib in Patients With Advanced Solid Tumors and Hematological Malignancies Characterized by Genetic Abnormalities of Anaplastic Lymphoma Kinase (ALK)
Brief Title: Ceritinib Rare Indications Study in ALK+ Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378A2407
Record Dates: First submitted 2015-05-29; First posted 2015-06-08 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Tumors With Aberrations in ALK; Anaplastic Large Cell Lymphoma; Inflammatory Myofibroblastic Tumor; Glioblastoma
Keywords: ALK; GBM; hematological malignancy; anaplastic lymphoma kinase; glioblastoma; anaplastic large cell lymphoma; IMT; inflammatory myofibroblastic tumor
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Granuloma, Plasma Cell; Glioblastoma; Hematologic Neoplasms | interventions — ceritinib

STUDY DESIGN:
Intervention Model Description: Depending on the tumor type, subjects were to be enrolled into one of the following parallel arms: ALCL (anaplastic large cell lymphoma); IMT (inflammatory myofibroblastic tumor); glioblastoma (GBM), and any other ALK+ tumor. If there were 5 or more subjects of the same tumor type in the "Any other ALK+ tumor" arm, then a separate arm was to be opened for that specific tumor type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Inflammatory myofibroblastic tumor (IMT) (Experimental): Patients diagnosed with IMT with a confirmed translocation involving the ALK gene
  Interventions: Drug: Ceritinib (LDK378)
- Anaplastic large cell lymphoma (ALCL) (Experimental): Patients with a diagnosis of ALCL histologically or cytologically confirmed to be ALK-positive
  Interventions: Drug: Ceritinib (LDK378)
- Glioblastoma (GBM) (Experimental): Patients with GBM with a translocation involving the ALK gene
  Interventions: Drug: Ceritinib (LDK378)
- Any other ALK-positive tumor (Experimental): Patients with any other ALK-positive tumor. Patients in this arm included adenocarcinoma (n= 2), sarcoma (1) and other (2).
  Interventions: Drug: Ceritinib (LDK378)

INTERVENTIONS:
Drug: Ceritinib (LDK378) — Ceritinib was to be administered orally once daily at a dose of 750 mg (5 capsules of 150 mg) on a continuous dosing schedule. A complete treatment cycle was defined as 28 days of once daily continuous treatment with ceritinib.

SUMMARY:
This is Proof-of-Concept (POC) study to assess the preliminary antitumor activity and safety and tolerablity using ceritinib (LDK378) in the treatment of life threatening tumors that are characterized by ALK genetic alteration (and/or overexpression in some diseases).

ELIGIBILITY:
Inclusion Criteria:

* Patient has a histologically or cytologically confirmed diagnosis of ALK positive (ALK+) tumor other than Non-Small Cell Lung Cancer (NSCLC).
* Patient must provide an archival or fresh tumor tissue before the first dose of the study drug for ALK testing at a Novartis designated central laboratory.
* Patient has WHO Performance Status (PS) ≤ 2
* Patient must have received at least one line of prior systemic treatment for recurrent, locally advanced and/or metastatic disease, and may have discontinued for:

  * Disease progression as defined by RECIST 1.1 for solid tumors; by RANO for GBM and by Cheson assessment criteria for lymphoma, or
  * Intolerance described as any discontinuation due to an AE of any grade despite appropriate supportive treatment
* Patient has at least one measurable lesion as defined by appropriate guidelines. A lesion at a previously irradiated site may only be counted as a target lesion if there is clear sign of progression since the irradiation.
* Patient has received no chemotherapy, immunotherapy or stem cell therapy at least 4 weeks before starting ceritinib
* Radiotherapy and prior ALK inhibitors must be stopped at least 1 week prior to starting ceritinib
* Recovered from all toxicities related to prior anticancer therapies to grade ≤ 1 (Common Terminology Criteria for Adverse Events [CTCAE] v4.03).

Exclusion Criteria:

* Patient has ALK+lung cancer
* Patient with symptomatic CNS metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms.
* Patient with acute or chronic GI disease that may significantly alter the absorption of ceritinib.
* Patient with a history of pancreatitis or history of increased amylase or lipase that was due to pancreatic disease.
* Patient has history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis.
* Patient has clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months).
* Patient has evidence of active viral hepatitis, including Hepatitis A, B or C (testing for viral hepatitis is not mandatory).
* Patient has known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Novartis Investigative Site, Brno, Czech Republic, Czechia
- Novartis Investigative Site, Copenhagen, Denmark
- France (3):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Saint-Herblain Cédex
  - Novartis Investigative Site, Strasbourg
- Novartis Investigative Site, Tel Aviv, Israel
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Madrid, Spain
- Novartis Investigative Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A minimum of 10 and a maximum of 20 subjects were to be enrolled in each arm (tumor type)
Period: Overall Study
Arm/Group | Anaplastic Large Cell Lymphoma (ALCL) | Inflammatory Myofibroblastic Tumor (IMT) | Glioblastoma (GBM) | Any Other ALK-positive Tumor
Started | 1 | 4 | 12 | 5
Completed | 0 | 0 | 0 | 0
Not Completed | 1 | 4 | 12 | 5
Not completed — Progressive disease | 0 | 2 | 9 | 4
Not completed — Study terminated by sponsor | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anaplastic Large Cell Lymphoma (ALCL) | Inflammatory Myofibroblastic Tumor (IMT) | Glioblastoma (GBM) | Any Other ALK-positive Tumor | Total
Number analyzed (Participants) | 1 | 4 | 12 | 5 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 | 42.8 (19.41) | 49.3 (15.40) | 57.4 (14.64) | 49.3 (15.85)
Age, Customized [Count of Participants; unit: Participants]
  18 to <65 | 1 | 4 | 10 | 3 | 18
  65 to <=75 | 0 | 0 | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 6 | 1 | 11
  Male | 0 | 1 | 6 | 4 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 0 | 1 | 10 | 2 | 13
  Asian | 1 | 1 | 1 | 3 | 6
  Other | 0 | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR) Based on Investigator Assessments for Participants With at Least 16 Weeks of Treatment
Description: The DCR is defined as the percentage of patients with complete response (CR), partial response (PR) or stable disease (SD) at 16 weeks from the start of ceritinib treatment. The assessment criteria are: Solid Tumors (RECIST 1.1., Response Evaluation Criteria in Solid Tumors); GBM (RECIST 1.1 and RANO, Response Evaluation in Neuro-Oncology); Hematologic tumors (Cheson).
Time Frame: Baseline up to approximately 16 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anaplastic Large Cell Lymphoma (ALCL) | Inflammatory Myofibroblastic Tumor (IMT) | Glioblastoma (GBM) | Any Other ALK-positive Tumor
Number analyzed (Participants) | 1 | 4 | 12 | 5
percentage of participants | 100.00 [2.5 to 100.0] | 75.00 [19.4 to 99.4] | 0.0 [0.0 to 26.5] | 40.0 [5.3 to 85.3]

2. Secondary Outcome: Overall Response Rate (ORR) Per Investigator Assessment
Description: ORR is defined as the percentage of patients with best overall response of complete response (CR) or partial response (PR) based on local assessment according to RECIST 1.1, RANO or Cheson hematological criteria.
Time Frame: Baseline, every 8 weeks until disease progression or end of treatment, whichever came first assessed up to approximately 84 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anaplastic Large Cell Lymphoma (ALCL) | Inflammatory Myofibroblastic Tumor (IMT) | Glioblastoma (GBM) | Any Other ALK-positive Tumor
Number analyzed (Participants) | 1 | 4 | 12 | 5
percentage of participants | 100.0 [2.5 to 100.0] | 75.0 [19.4 to 99.4] | 0.0 [0 to 26.5] | 0.0 [0.0 to 52.2]

3. Secondary Outcome: Duration of Response (DOR) Per Investigator Assessment
Description: DOR is defined as the time from date of first documented CR or PR to date of first documented disease progression or death due to any cause
Time Frame: Baseline, every 8 weeks until disease progression or end of treatment, whichever came first, assessed up to approximately 84 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Glioblastomia (GBM): Patients with GBM with a translocation involving the ALK gene
Arm/Group | Anaplastic Large Cell Lymphoma (ALCL) | Inflammatory Myofibroblastic Tumor (IMT) | Glioblastomia (GBM) | Any Other ALK-positive Tumor
Number analyzed (Participants) | 1 | 3 | 12 | 5
weeks | NA [NA to NA] — Median was not reached for DOR therefore Confidence Interval was not estimable | NA [3.0 to NA] — Median was not reached for DOR | NA [NA to NA] — No participants experienced CR or PR for this cohort | NA [NA to NA] — No participants experienced CR or PR for this cohort

4. Secondary Outcome: Time to Response (TTR) Per Investigator Assessment
Description: TTR is defined as the time from date of the first dose to date of first documented response (CR or PR)
Time Frame: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Anaplastic Large Cell Lymphoma (ALCL) | Inflammatory Myofibroblastic Tumor (IMT) | Glioblastoma (GBM) | Any Other ALK-positive Tumor
Number analyzed (Participants) | 1 | 4 | 12 | 5
weeks | 7.1 [NA to NA] — Confidence Interval was not estimable | 16.4 [6.3 to NA] — Upper Confidence Interval was not estimable | NA [NA to NA] — No participants experienced CR or PR for this cohort | NA [NA to NA] — No participants experienced CR or PR for this cohort

5. Secondary Outcome: Progression Free Survival (PFS) Per Investigator Assessments
Description: PFS is defined as the time from the date of first dose of ceritinib to the date of first documented disease progression or death from any cause
Time Frame: Baseline, every 8 weeks until disease progression or death from any cause, assessed for up to approximately 84 weeks
Population: no participants met definition of PFS
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Anaplastic Large Cell Lymphoma (ALCL) | Inflammatory Myofibroblastic Tumor (IMT) | Glioblastoma (GBM) | Any Other ALK-positive Tumor
Number analyzed (Participants) | 0 | 2 | 9 | 5
weeks |  | NA [3.7 to NA] — Median and upper CI were not estimable | 1.7 [1.1 to 2.7] | 1.7 [1.6 to 5.1]

6. Secondary Outcome: Percent of Participant Deaths During Treatment and Follow-up
Description: Deaths due to any cause during treatment and 30 day follow-up
Time Frame: Baseline up to approximately 84 weeks
Population: There were no deaths in the ALCL and IMT arms
Measure: Number; unit: percent of participants
Arm/Group | Anaplastic Large Cell Lymphoma (ALCL) | Inflammatory Myofibroblastic Tumor (IMT) | Glioblastoma (GBM) | Any Other ALK-positive Tumor
Number analyzed (Participants) | 1 | 4 | 12 | 5
percent of participants | 0.0 | 0.0 | 25.0 | 20.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of 84 weeks
Description: Any sign or symptom that occured during the study treatment plus 30 days post treatment
Groups:
- Anaplastic Large Cell Lymphoma: Anaplastic Large Cell Lymphoma
- Inflammatory Myofibroblastic Tumor: Inflammatory Myofibroblastic Tumor
- Glioblastoma: Glioblastoma
- Any Other ALK+ Tumor: Any other ALK+ tumor
- All Subjects: All Subjects
Arm/Group | Anaplastic Large Cell Lymphoma | Inflammatory Myofibroblastic Tumor | Glioblastoma | Any Other ALK+ Tumor | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/4 | 3/12 | 1/5 | 4/22
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/4 | 10/12 | 4/5 | 16/22
Other Adverse Events (participants affected / at risk) | 1/1 | 4/4 | 12/12 | 5/5 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anaplastic Large Cell Lymphoma (N=1) | Inflammatory Myofibroblastic Tumor (N=4) | Glioblastoma (N=12) | Any Other ALK+ Tumor (N=5) | All Subjects (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 2 | 4
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 2 | 0 | 2
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Hypersomnia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Paraneoplastic pemphigus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anaplastic Large Cell Lymphoma (N=1) | Inflammatory Myofibroblastic Tumor (N=4) | Glioblastoma (N=12) | Any Other ALK+ Tumor (N=5) | All Subjects (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 3 | 5
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 2 | 5
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 7 | 2 | 13
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 6 | 3 | 13
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2 | 4 | 4 | 11
Asthenia (General disorders) | 0 | 0 | 1 | 4 | 5
Fatigue (General disorders) | 0 | 1 | 5 | 0 | 6
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 3 | 0 | 3
Pain (General disorders) | 0 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Candiduria (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Genital herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 2
Uterine infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 3 | 2 | 1 | 7
Amylase increased (Investigations) | 0 | 2 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 0 | 1 | 5
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 0 | 1 | 4
Blood bilirubin abnormal (Investigations) | 0 | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 2 | 0 | 0 | 2
Creatinine renal clearance increased (Investigations) | 0 | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 0 | 1 | 4
Lipase increased (Investigations) | 0 | 1 | 0 | 1 | 2
Weight decreased (Investigations) | 0 | 0 | 1 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 2 | 0 | 2
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 3 | 0 | 3
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 2 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 3
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-11-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT02465528/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT02465528/SAP_001.pdf